CLINICAL TRIAL: NCT04744896
Title: Effects Of Combined Cryolipolysis And High Intensity Interval Training On Insulin Resistance And Body Composition In Polycystic Ovarian Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Miral Saleh Mohamed, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EHCIBPP
Record Dates: First submitted 2021-02-03; First posted 2021-02-09 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Polycystic Ovary Syndrome; Hyperinsulinism
Keywords: pco
MeSH Terms: conditions — Polycystic Ovary Syndrome; Hyperinsulinism

STUDY DESIGN:
Intervention Model Description: cryolipolysis treadmill cryolipolysis + treadmill
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cryolipolysis (Experimental): 3max cool shaping device is administered 3 times for each patient, one session every 6 weeks, each session is 40 minutes.
  Interventions: Device: cryolipolysis(3 max cool shaping)
- treadmill (Experimental): aerobic training in form of high intensity interval training, three times per week for 3 weeks by treadmill(jkexer focus 8020A) each session is for 20 minutes.
  Interventions: Device: Treadmill (jkexer focus 8020A)
- treadmill+cryolipolysis (Active Comparator): aerobic training 3 times per week and cryolipolysis once every 6 weeks
  Interventions: Device: cryolipolysis(3 max cool shaping); Device: Treadmill (jkexer focus 8020A)

INTERVENTIONS:
Device: cryolipolysis(3 max cool shaping) — cryolioplysis applied over abdomen area
  Arms: cryolipolysis; treadmill+cryolipolysis
Device: Treadmill (jkexer focus 8020A) — aerobic training ( high intensity interval training)
  Arms: treadmill; treadmill+cryolipolysis

SUMMARY:
this study will be carried to investigate the effect of cryolipolysis and high intensity interval training on insulin resistance and body composition in pco women

DETAILED DESCRIPTION:
This study will be carried out on ninety females with polycystic ovarian syndrome (PCOS)l. Their age ranges from 17-28 years, body mass index 25-30 Kg/m2. They experience hyperandrogenism and hyperinsulinemia.

PCOS females will be randomly assigned into three equal groups: group (A) consists of 30 women who receive cryolipolysis and group (B) consists of 30 women who receive high intensity interval training and group (C) receive both

ELIGIBILITY:
Inclusion Criteria:

* women diagnosed with polycystic ovarian syndrome
* age ranges from 17-28 years
* body mass index ranges 25-30 Kg/m2

Exclusion Criteria:

* Diabetic patients.
* Women with BMI>30
* Women having circulatory dysfunction.
* Women with respiratory or cardiac disease
* liver disease.
* Skin disease .
* Previous abdominal or uterine surgery
* any medications affecting hormones
* any physical impairments
* Physical impairment

Ages: 17 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
HOMA IR | 3 months
  blood test
weight | up to 3 months
  anthropometric measure measured in kilogram (kg)
fat percentage | up to 3 months
  overall body fat percentage measured by body fat analyzer in percentage (%)

SECONDARY OUTCOMES:
waist circumference | up to 3 months
  anthropometric measurement measured in centimeter (cm)

CONTACTS AND LOCATIONS:
Overall Officials: amal mo youssef, phd, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided